CLINICAL TRIAL: NCT07188155
Title: Adapting Exposure Therapy to Target Anxiety About Weight Gain in Adolescents With Anorexia Nervosa
Brief Title: Adapting Exposure for Adolescent AN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jamal Essayli, Assistant Professor of Pediatrics and Psychiatry & Behavioral Health, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27028
Record Dates: First submitted 2025-09-13; First posted 2025-09-23 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; exposure therapy; adolescents
MeSH Terms: conditions — Anorexia Nervosa | interventions — Implosive Therapy; Appetite Depressants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposure Therapy for AN (Exp-AN) (Experimental): Exp-AN aims to target anxiety about weight gain by helping participants identify their specific feared consequences of weight gain (e.g., "I will permanently hate myself if I gain weight"), and combining in vivo (i.e., in real life) and imaginal (i.e., mental) exposure exercises to address these fears. Exp-AN consists of four core modules: (1) Treatment Rationale and Psychoeducation; (2) In-Session Weight Exposure; (3) Planning, Conducting, and Reviewing Exposures; and (4) Relapse Prevention.
  Interventions: Behavioral: Exposure Therapy for Anorexia (Exp-AN)

INTERVENTIONS:
Behavioral: Exposure Therapy for Anorexia (Exp-AN) — Exp-AN is specifically designed to target anxiety about weight gain. Exp-AN helps participants identify their specific feared consequences of weight gain (e.g., "I will permanently hate myself if I gain weight"), and combines in vivo (i.e., in real life) and imaginal (i.e., mental) exposure exercises to address these fears.

SUMMARY:
This pilot study is evaluating Exposure Therapy (Exp-AN) as a virtual treatment for adolescents (ages 14 - 17 years) with anorexia nervosa (AN) recruited from eating disorder clinic waitlists and clinician referrals at the Penn State Milton S. Hershey Medical Center and the University of California, San Francisco (UCSF) (8 participants per site). Adolescents who agree to take part in this study will receive 20 free virtual 40-60 minute weekly Exp-AN sessions at an outpatient level of care. Exp-AN for adolescents will combine individual virtual session time (35-50 min) with parent involvement (10-25 min). Parents will serve as "collaborators," supporting skill development, exposure completion, and treatment goal achievement. Exp-AN sessions will focus on helping participants overcome anxiety about weight gain by encouraging them to do challenging things that increase anxiety in the short term but help them better tolerate anxiety over the long term. Participants will be asked to complete a clinical interview, questionnaires, and labs and vitals testing before they begin the study. Adolescents will also complete questionnaires and participate in 15-min semi-structured interviews, while parents/caregivers will complete separate parallel interviews, at: mid-treatment, end-of-treatment, and 3-month follow-up. To ensure that all participants are receiving the same type of therapy, they will not be able to have any concurrent psychotherapy while receiving this treatment (other forms of care including dieticians, nutritionists, and psychiatrists are allowed).

Exp-AN is designed to target anxiety about weight gain. Exp-AN includes education about the effects of undereating; the importance of overcoming anxiety about weight gain; in-session weight exposures (e.g., stepping on a scale while reading a script describing fears about weight gain); creating a meal plan to help improve eating; reviewing eating behaviors over the past week; conducting in-session and between-session exposures that help participants face fears related to weight gain; and relapse prevention.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of anorexia nervosa (AN)
* English speaking
* Mentally stable for an outpatient level of care
* Living with at least one parent/caregiver
* Less than or equal to 90% of expected body weight

Exclusion Criteria:

* Younger than 14 years old or older than 17 years old
* Has a current psychotherapist and not open to pausing treatment for the duration of the study
* Has a diagnosis of bulimia nervosa or binge-eating disorder
* Acutely suicidal
* Pregnant
* Meets DSM-5 criteria for a psychotic disorder and/or has an intellectual disability
* Non-English speaking

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Examination - Self-Report Questionnaire (EDE-Q) | Baseline, Mid-Treatment, End-of-Treatment, 3-Month-Follow-Up
  The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-report questionnaire. It was designed to assess the range, frequency, and severity of behaviors associated with a diagnosis of an eating disorder. A global score is obtained by summing the four subscales scores (ranging from 0-6) and dividing the total by the number of subscales (4). The score of items are calculated and range from 0 to 6. The higher score indicate greater ED symptoms.
Fear of Food Measure (FOFM) | Baseline, Mid-Treatment, End-of-Treatment, 3-Month-Follow-Up
  The Fear of Food Measure (FORM) is a 23-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. Each item is scored on a 1-7 scale. The questionnaire range from 23 to 161 meaning 23: no fear of food and 161 meaning severe fear of food.
Body Shape Questionnaire (BSQ) | Baseline, Mid-Treatment, End-of-Treatment, 3-Month-Follow-Up
  The BSQ is a self-reported measurement of the body shape concerns typical of bulimia nervosa and anorexia nervosa. The questionnaire has 34 items scored from 0 to 6 points (least and most impaired, respectively), with the sum of the questions giving a range from 0 to 204. The higher score indicates greater concerns about body shape.
Clinical Impairment Assessment (CIA) | Baseline, Mid-Treatment, End-of-Treatment, 3-Month-Follow-Up
  The Clinical Impairment Assessment Questionnaire (CIA) is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features and focuses on the past 28 days. The 16 items cover impairment in domains of life that are typically affected by eating disorder psychopathology: mood and self-perception, cognitive functioning, interpersonal functioning, and work performance. The responses are scored 0,1,2 and 3, with a higher rating indicating a higher level of impairment. The total range is between 0 and 48.
Eating Disorder Fear Questionnaire (EDFQ) | Baseline, Sessions 1-20, 3-Month-Follow-Up
  The Eating Disorder Fear Questionnaire (EDFQ) is a 20-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. The response range between 1 to 7 with a total range of 20 to 140. The higher rating indicates a higher severe impairment.
Weight Gain Anxiety Questionnaire | Baseline, Sessions 1-20, 3-Month-Follow-Up
  The Weight Gain Anxiety Questionnaire is a 12-item self-report questionnaire that targets anxiety about weight gain. The scores are measured on a 0-100 scale, with the higher the score indicating more distress about weight gain, with the exception for question 2 which is reverse scored.
Eating Anxiety Questionnaire | Baseline, Sessions 1-20, 3-Month-Follow-Up
  The Eating Gain Anxiety Questionnaire is a 14-item self-report questionnaire that targets anxiety about eating fear foods. The scores are measured on a 0-100 scale, with the higher the score indicating more distress about eating fear foods, with the exception for question 2 which is reverse scored.
Patient Health Questionnaire-9 (PHQ-9) | Baseline, Mid-Treatment, End-of-Treatment, 3-Month-Follow-Up
  The Patient Health Questionnaire-9 is a 9-item self-report questionnaire that targets depressive symptoms. The scores range from 0-27, with higher scores indicating a higher level of depression.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline, Mid-Treatment, End-of-Treatment, 3-Month-Follow-Up
  The Generalized Anxiety Disorder-7 is a 7-item self-report questionnaire that targets anxiety symptoms. The scores range from 0 to 21, with higher scores indicating higher levels of anxiety.
Eating Disorder Examination - Self-Report Questionnaire Parent Version 1.5 (PEDE-Q) | Baseline, Mid-Treatment, End-of-Treatment, 3-Month-Follow-Up
  Eating Disorder Examination - Self-Report Questionnaire Parent Version 1.5 (PEDE-Q) is a 29-item self-report questionnaire. It is intended to be completed by the parent of a child with an eating disorder targeting the parent's perspective of their child's eating disorder. It was designed to assess the range, frequency, and severity of behaviors associated with a diagnosis of an eating disorder. A global score is obtained by summing the four subscales scores (ranging from 0-6) and dividing the total by the number of subscales (4). The score of items are calculated and range from 0 to 6. The higher scores indicate greater perceived child's ED symptoms.
Parent vs Eating Disorder Scale (PVED) | Baseline, Mid-Treatment, End-of-Treatment, 3-Month-Follow-Up
  The Parent vs Eating Disorder Scale (PVED) is a 7-item self-report questionnaire that examines parents' opinions on parent involvement in the treatment of their child's eating disorder. Higher scores indicate higher agreement with the statements, and lower scores indicate lower agreement with the statements. Scores range from 1 (strongly disagree) - 5 (strongly agree).
Percent of Expected Body Weight (EBW) | Baseline, Mid-Treatment, End-of-Treatment, 3-Month-Follow-Up
  We will measure the participants' weight using a wireless smart scale.

SECONDARY OUTCOMES:
Treatment Acceptability Questionnaire | Baseline, Mid-Treatment, End-of-Treatment, 3-Month-Follow-Up
  The Treatment Acceptability Questionnaire is a 10-item self-report questionnaire. It examines the participants' perspective on the modules in the exposure therapy. The response range between 1 to 7, with a total range of 10 to 70. The higher rating indicates a higher rating of treatment acceptability.
Recruitment | Through study completion, an average of 2 years
  We will measure recruitment by calculating the percentage of eligible participants approached who consent to the study. The higher the percentage, the more successful we were with recruiting for the study.
Retention | Through study completion, an average of 2 years
  We will measure the percent of participants who complete the study by calculating the percentage of participants that complete the three-month follow-up. The higher the percentage, the more participants completed the study.
Engagement | Through study completion, an average of 2 years
  We will measure participant engagement by calculating the number of sessions participants attend out of 20 total sessions. The higher the number of sessions attended, the more participant engagement in the study.
Treatment Fidelity | Through study completion, an average of 2 years
  We will measure the therapists' adherence to the protocol by completing a treatment adherence measure that measures the study interventionists' adherence to the protocol. The higher the treatment adherence measure, the more the study interventionists adhered to the protocol.

IPD SHARING:
Plan to Share IPD: Undecided